CLINICAL TRIAL: NCT03773497
Title: Bioavailability of Phytonutrients From Novel Preparations of Broccoli
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Craig Charron, Research Molecular Biologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HS63 - Broccoli Snack Study
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Common snack combination (Other): Subjects will consume a self-chosen, low-carotenoid diet, and on the first day, with breakfast, will consume a snack of a combination of common snack foods (pretzels, potato chips, and popcorn).
  Interventions: Other: Common Snack Combination
- Cheese broccoli (Other): Subjects will consume a self-chosen, low-carotenoid diet, and on the first day, with breakfast, will consume a snack of oven-roasted, freeze-dried, cheese flavored broccoli.
  Interventions: Other: Cheesy Broccoli Snack
- Cheese broccoli with Daikon radish powder (Other): Subjects will consume a self-chosen, low-carotenoid diet, and on the first day, with breakfast, will consume a snack of oven-roasted, freeze-dried, cheese flavored broccoli with Daikon radish powder.
  Interventions: Other: Cheesy Broccoli with Daikon Radish Snack
- Uncooked broccoli with ranch-type dip (Other): Subjects will consume a self-chosen, low-carotenoid diet, and on the first day, with breakfast, will consume a snack of uncooked, freeze-dried broccoli with ranch-type dip.
  Interventions: Other: Uncooked Broccoli Snack

INTERVENTIONS:
Other: Common Snack Combination — Combination of Chips, Pretzels, and Popcorn.
  Arms: Common snack combination
Other: Cheesy Broccoli Snack — Oven-roasted, freeze-dried, cheese flavored broccoli
  Arms: Cheese broccoli
Other: Cheesy Broccoli with Daikon Radish Snack — Oven-roasted, freeze-dried, cheese flavored broccoli with Daikon radish powder
  Arms: Cheese broccoli with Daikon radish powder
Other: Uncooked Broccoli Snack — Uncooked, freeze-dried broccoli with ranch-type dip
  Arms: Uncooked broccoli with ranch-type dip

SUMMARY:
The primary objective of this study is to determine the effects of different methods of broccoli preparation on levels of urinary glucosinolate metabolites. The secondary objective is to determine the effects of different methods of broccoli preparation on levels of plasma carotenoids.

DETAILED DESCRIPTION:
Consumption of Brassica vegetables (which include broccoli, cabbage, and kale) is inversely associated with the incidence of several cancers, including cancers of the lung, stomach, liver, colon, rectum, breast, endometrium, and ovaries. Brassica vegetables are a good source of many nutrients including glucosinolates and carotenoids. Glucosinolates are sulfur-containing compounds that are converted to bioactive metabolites by an enzyme called myrosinase, which is released when the vesicles containing myrosinase are ruptured by chewing or cutting. These bioactive compounds are considered to be active agents for cancer prevention. Their ability to reduce risk of cancer may derive in part from their ability to modulate foreign-substance metabolizing enzymes, which include enzymes called Phase I cytochrome P450s and Phase II enzymes. Carotenoids may also have a role in cancer prevention and other health benefits including reducing age-related macular degeneration, and therefore merit research to reveal factors that affect their presence in the body.

The primary aim of this study is to investigate how various preparations of broccoli impact levels of these healthful nutrients in humans.

ELIGIBILITY:
Inclusion Criteria:

* Between 21 and 75 years old at beginning of study

Exclusion Criteria:

* Pregnant, lactating, or intending to become pregnant during the study period
* Women who have given birth during the previous 12 months
* Presence of kidney disease, liver disease, gout, certain cancers, gastrointestinal disease, hyperthyroidism, untreated or unstable hypothyroidism, pancreatic disease, other metabolic diseases, or malabsorption syndromes requiring special diets
* History of certain cancers within last 3 years
* Known allergy or intolerance to Brassica vegetables
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low-fat diets, high-protein diets)
* Colonoscopy during three weeks prior to start of study
* Unwillingness to abstain from probiotics or vitamin, mineral, herbal and glucosinolate/isothiocyanate supplements for two weeks prior to the study and during the study
* Use of tobacco products within 6 months preceding study
* Crohn's disease or diverticulitis
* Suspected or known strictures, fistulas or physiological/mechanical GI obstruction
* Use of certain medications (prescription or over-the-counter) that may interfere with the study objectives
* Type 2 diabetes requiring the use of diabetes pills, insulin, or non-insulin shots
* Fasting glucose greater than or equal to 126 mg/dL
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current treatment for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Glucosinolate Metabolites will be measured | Day 1
  Urine will be analyzed for glucosinolate metabolites
Glucosinolate Metabolites will be measured | Day 22
  Urine will be analyzed for glucosinolate metabolites
Glucosinolate Metabolites will be measured | Day 43
  Urine will be analyzed for glucosinolate metabolites
Glucosinolate Metabolites will be measured | Day 64
  Urine will be analyzed for glucosinolate metabolites

SECONDARY OUTCOMES:
Carotenoids will be measured | Days 1, 2, 3, 4, 11, 22, 23, 24, 25, 32, 43, 44, 45, 46, 53, 64, 65, 66, 67, 74
  Carotenoids will be extracted from plasma

CONTACTS AND LOCATIONS:
Locations (1):
- USDA-ARS Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No